CLINICAL TRIAL: NCT02537236
Title: Efficacy and Safety of Fish Oil (Omega-3 Fatty Acid) Supplementation With Therapeutic Lifestyle Changes Diet Associated With Lipidic Profile in HIV-positive Patients With Antiretroviral Therapy.
Brief Title: Omega-3 Supplementation in HIV Patients With Therapeutic Lifestyle Change Diet.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Alejandro Gonzalez-Ojeda, MD., Ph.D., F.A.C.S., Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: omega-3-HIV/2009
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: Omega-3 Fatty Acids; Therapeutic Lifestyle Changes; Human Immunodeficiency Virus; Cardiac Risk; Dyslipidemia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Dyslipidemias | interventions — Fatty Acids, Omega-3; Eicosapentaenoic Acid; Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group one (Experimental): 20 subjects received Therapeutic Lifestyle Changes diet more 1.05 grams of fish oil omega 3 fatty acids
  Interventions: Dietary Supplement: Omega-3 fatty acid supplementation with fish oil and TLC nutritional intervention.
- Group two (Active Comparator): 20 subjects received conventional diet more 1.05 grams of fish oil omega 3 fatty acids
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Group three (Experimental): 20 subjects received Therapeutic Lifestyle Changes diet more 2.10 grams of fish oil omega 3 fatty acids.
  Interventions: Dietary Supplement: Omega-3 fatty acid supplementation with fish oil and TLC nutritional intervention.
- Group four (Active Comparator): 20 subjects received conventional diet more 2.10 grams of fish oil omega 3 fatty acids
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Group five (Placebo Comparator): 20 subjects, control group received conventional diet.
  Interventions: Behavioral: TLC nutritional intervention

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — Omega-3 fatty acid supplementation with fish oil.
  Other Names: eicosapentaenoic acid; docosahexaenoic acid
  Arms: Group four; Group two
Behavioral: TLC nutritional intervention — nutritional orientation.
  Arms: Group five
Dietary Supplement: Omega-3 fatty acid supplementation with fish oil and TLC nutritional intervention. — Omega 3 fatty acid supplementation with fish oil and nutritional counseling of TLC diet.
  Arms: Group one; Group three

SUMMARY:
The positive patients to the Human Immunodeficiency Virus (HIV) with Highly Active Antiretroviral Therapy (HAART) present multiple alterations in their corporal composition and dyslipidemia, wich increase the cardiovascular risk.

The investigators evaluated the efficiency of the combination of fish oil omega 3 fatty acids to different doses with the Therapeutic Lifestyle Changes (TLC) diet of the National Cholesterol Education Program on the profile of lipids and the corporal weight in patients with HIV treated with HAART.

DETAILED DESCRIPTION:
The infection by Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS), is a chronic condition transmissible and progressive type of viral cause, in which a link is very different between host and virus, which ultimately influences the appearance of opportunistic morbid processes or rare tumors, or both1.

With a prevalence of 3 cases for every 1000 people from 15 to 49 years, Mexico ranks 16th place in the prevalence of HIV/AIDS in adults in Latin America2.

The state of Jalisco, México, occupies the fourth place in terms of positive cases of HIV-AIDS, in this same plane, the municipalities of Guadalajara, Zapopan, Tlaquepaque and Puerto Vallarta in Jalisco, represent the main populations with the highest number of positive cases by HIV-AIDS.

The HIV positive individuals with Highly Active Antiretroviral Therapy (HAART) or without treatment are facing numerous challenges in terms of management of their health; some of the most disturbing changes are visible in the shape and appearance of the body. In most cases this anatomical changes come accompanied by alterations in biochemical indicators: lipid levels (cholesterol and triglycerides) and insulin resistance4.These adverse effects may have important clinical implications, such as severe lactic acidosis, coronary artery disease and acute pancreatitis5.

In patients with HIV and HAART has published an incidence of hypercholesterolemia and hypertriglyceridemia between 5 and 90% depending on the series, although the true incidence is yet to be determined6. Pharmacological interventions with statins or fibrates in patients infected with HIV are limited partially due to the drug interactions and increase in the frequency of adverse effects7.

Therefore, it is necessary to investigate new alternatives for the management of dyslipidemia in patients infected with HIV with HAART through changes in diet and supplements of fish oil omega 3 fatty acids.

Methods Patients: The investigators enrolled 100 Patients positive to Human Immunodeficiency Virus or Acquired Immunodeficiency Syndrome, and had been receiving ≥2 Highly Active Antiretroviral Therapy, and with diagnostic of dislipidemia according the Mexican Official Standard Norms of 2002, for the prevention, treatment and control of dyslipidemias8.

All the patients were active in the SMART database from HIV/AIDS department of the Civil Hospital in Guadalajara "Fray Antonio Alcalde". Patients were excluded for intolerance or allergy to fish, patients that use or have used in the last 6 weeks supplements or drugs that modify lipids.

Study design During the period from January 2010 to July 2011, was carried out the study with the authorization of the ethics committee of the Civil Hospital in Guadalajara "Fray Antonio Alcalde".

Our subjects were assigned to 5 intervention groups: Groups one= 20 subjects received Therapeutic Lifestyle Changes diet more 1.05 grams of Fatty Acid omega 3. Groups two= 20 subjects received conventional diet more 1.05 grams of Fatty Acid omega three. Groups 3=20 subjects received Therapeutic Lifestyle Changes diet more 2.10 grams of Fatty Acid omega 3. Groups four=20 subjects received conventional diet more 2.10 grams of Fatty Acid omega 3. Groups five= 20 subjects, control group received conventional diet.

The subject assigned to group one and three with TLC diet, received advice from the nutritionist in week 4 and 12 to encourage the consumption of the capsules of omega 3 fatty acids, in addition offered general recommendations to consume dietary fiber and fluids.

The subject assigned to groups two and four with conventional diet, received advice from the nutritionist in the week 4 and 12 to encourage the consumption of the capsules of omega 3 fatty acids without the assistance of special diet.

The requirements of energy and macronutrients were identified in the patients of group one and three.

None of the subjects received advice on the physical activity that could perform.

Statistical analysis

The main objective of this study was to compare the changes in fasting levels of triglycerides (TG), total cholesterol (TC), high density cholesterol (HD-C), low density cholesterol (LD-C), very low density cholesterol (VLD-C), the body weight and body mass index (BMI) against the week 4 and 12.

The safety and tolerability of the study medication were also secondary outcomes.

Statistical analysis was carried out starting with the Kolmogorov-Smirnov test to identify the distribution of variables, then identify the type of distribution of each variable, is continuous with the descriptive statistical analysis for variables with abnormal distribution -non-parametric, with measures of central tendency and dispersion as: the median distance and interquartiles and variables with normal distribution - parametric- :the mean and standard deviation.

Inferential analysis to the intra-group used the Wilcoxon test and Friedman. For the inferential analysis between groups was implemented in the variables of non-normal distribution, the Kruskal-Wallis test; and for variables with normal distribution was used the one-way ANOVA test. Differences were considered statistically significant when the p value was <0.05 .

The data were processed using the statistical package No.18.0 and are presented in tables and graphics.

ELIGIBILITY:
Inclusion Criteria:

* Patients positive to Human Immunodeficiency Virus or Acquired Immunodeficiency Syndrome
* Patients older than 18 years positive to HIV/AIDS with HAART
* Patients who agreed to sign consent under written information
* Patients that had some type of dyslipidemia according the Mexican Norms of 2002.

Exclusion Criteria:

* Patient with mouth non-permeable
* Patients with intolerance or allergy to fish oil
* Patient record in the database SMART but inactive.
* Patients who use or have used in the last 6 weeks food supplements that modify lipids.
* Patient who have not attended two of the four set appointments for valuation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Triglycerides (TG) | At baseline
  Serum TG measured at baseline, before initiating treatment.
Total cholesterol (TC) | At baseline
  Serum TC measured at baseline, before initiating treatment.
High density cholesterol (HD-C) | At baseline
  Serum HD-C measured at baseline, before initiating treatment
Low density cholesterol (LD-C) | At baseline
  Serum LD-C measured at baseline, before initiating treatment
Very low density cholesterol (VLD-C) | At baseline
  Serum VLD-C measured at baseline, before initiating treatment
Body weight | At baseline
  Total weight before initiating treatment.
Body mass index (BMI) | At baseline
  BMI obtained before initiating treatment
TG 4 | At week four of treatment
  Serum TG measured at week four of treatment.
TC 4 | At week four of treatment
  Serum TC measured at week four of treatment.
HD-C 4 | At week four of treatment
  Serum HD-C measured at week four of treatment.
LD-C 4 | At week four of treatment
  Serum LD-C measured at week four of treatment.
VLD-C 4 | At week four of treatment
  Serum VLD-C measured at week four of treatment.
Weight 4 | At week four of treatment
  Total weight before at week four of treatment.
BMI 4 | At week four of treatment
  BMI obtained at week four of treatment
TG 12 | At week twelve of treatment
  Serum TG measured at week four of treatment.
TC 12 | At week twelve of treatment
  Total serum TG measured at week twelve of treatment
HD-C 12 | At week twelve of treatment
  Serum HD-C measured at week twelve of treatment
LD-C 12 | At week twelve of treatment
  Serum LD-C measured at week twelve of treatment
VLD-C 12 | At week twelve of treatment
  Serum VLD-C measured at week twelve of treatment
Weight 12 | At week twelve of treatment
  Total weight before at week twelve of treatment.
BMI 12 | At week twelve of treatment
  BMI obtained at week twelve of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro González-Ojeda, MD. PhD. F.A.C.S., Study Director — Instituto Mexicano del Seguro Social

REFERENCES:
- [Background] Carr A, Samaras K, Burton S, Law M, Freund J, Chisholm DJ, Cooper DA. A syndrome of peripheral lipodystrophy, hyperlipidaemia and insulin resistance in patients receiving HIV protease inhibitors. AIDS. 1998 May 7;12(7):F51-8. doi: 10.1097/00002030-199807000-00003. PMID 9619798
- [Background] Mulligan K, Grunfeld C, Tai VW, Algren H, Pang M, Chernoff DN, Lo JC, Schambelan M. Hyperlipidemia and insulin resistance are induced by protease inhibitors independent of changes in body composition in patients with HIV infection. J Acquir Immune Defic Syndr. 2000 Jan 1;23(1):35-43. doi: 10.1097/00126334-200001010-00005. PMID 10708054
- [Background] Wohl DA, Tien HC, Busby M, Cunningham C, Macintosh B, Napravnik S, Danan E, Donovan K, Hossenipour M, Simpson RJ Jr. Randomized study of the safety and efficacy of fish oil (omega-3 fatty acid) supplementation with dietary and exercise counseling for the treatment of antiretroviral therapy-associated hypertriglyceridemia. Clin Infect Dis. 2005 Nov 15;41(10):1498-504. doi: 10.1086/497273. Epub 2005 Oct 11. PMID 16231263